CLINICAL TRIAL: NCT03285451
Title: Correlative Analysis of Upper Airway Collapse in Sleep Endoscope and Submental Ultrasound
Brief Title: Drug Induced Submental Ultrasound in Obstructive Sleep Apnea Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 06-X07-017
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Submental ultrasound, Obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: submental ultrasonography — Submental ultrasound, the noninvasive and convenient tool, has been widely applied to measure the tongue base thickness in patients with obstructive sleep apnea, so as to predict the severity and relationship with upper airway collapse.

SUMMARY:
In this study, submental ultrasound during awake and simultaneous under Drug-induced sleep endoscopy is applied in the diagnostic workup of obstructive sleep apnea patients. The aim is to assess the tongue base thickness during awake and sleep with different head positions. By correlation with Drug-induced sleep endoscopy findings, more parameters could be used for evaluation and management of upper airway collapse in obstructive sleep apnea patients.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a syndrome characterized by recurrent episodes of apnea and hypopnea during sleep that are caused by repetitive upper airway (UA) collapse and often result in decreased blood oxygen levels and arousal from sleep. Successful treatment lies in precise mapping the site of airway narrowing.

Drug-induced sleep endoscopy (DISE) is a well described modality to mimic the dynamic change of UA in OSA patients during natural sleep. Nevertheless, the tongue base thickness (TBT), one of the important anatomic factors in OSA, is hard to evaluate under this method. Recently, submental ultrasound (US), the noninvasive and convenient tool, has been widely applied to measure the TBT in awake OSA patients, so as to predict the severity and relationship with UA collapse. However, few evidence has addressed the relationship between UA collapse and the TBT in different head positions, awake and sleep period In this study, submental US during awake and drug induced sleep period is applied in the diagnostic workup of OSA patients. By correlation with DISE findings, more parameters could be used for evaluation and management of upper airway collapse in OSA patients.

Key Words: Submental ultrasound, Obstructive sleep apnea, Drug-induced sleep endoscopy

ELIGIBILITY:
Inclusion Criteria:

* Obstructive sleep apnea patients, age between 20-70

Exclusion Criteria:

* severe heart, lung, liver, and kidney comorbidity propofol or dexmedetomidine allergies (albeit rare)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obstructive sleep apnea patients, age between 20-70 without severe heart, lung, liver, and kidney comorbidity or propofol or dexmedetomidine allergies
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
The value of drug induced sleep ultrasonography in patients with obstructive sleep apnea | May, 2017 to Aug, 2017
  In this study, we proposed a novel method, drug induced sleep ultrasonography (DISU), which was applied to measure the tongue base thickness in OSA patients during drug induced sleep, so as to further understand the impact of dynamic change of tongue base thickness in OSA patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Chin Lan, MD, Study Chair — Taipei Tzu Chi Hospita l Buddhist Tzu Chi Medical Foundation
Locations (1):
- Taipei Tzu Chi Hospital Buddhist Tzu Chi Medical Foundation, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No